CLINICAL TRIAL: NCT04297579
Title: Congenital Nevi in the Lower Limb in Children : Which Size Can be Afforded by a Simple Surgical Procedure ?
Brief Title: Congenital Naevi of Lower Limb in the Child
Acronym: NAEVUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0063
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Congenital Melanocytar Nevi in the Lower Limb
Keywords: congenital nevi; naevus; Congenital skin neoplasm; Reconstructive surgical procedures
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depending on its dimensions, it is difficult to predict if a congenital nevi of the lower limb can be surgically removed by a unique simple procedure or by a complex procedure (expander, skin graft etc..), with a good result.

This study retrospectively reviewed the practice of our team of surgeons depending on the size of the naevus to reveal a dimension threshold that can be used in the future to help to choose between a simple or a complex procedure.

DETAILED DESCRIPTION:
Retrospective study using medical file data only. No intervention nor phone call etc.. to the patients or their parents.

ELIGIBILITY:
Inclusion criteria:

- Child + congenital nevi in the lower limb + had removal surgery

Exclusion criteria:

- More than one congenital nevi in the lower limb.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children that had congenital nevi surgery removal, in the lower limb.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 1984-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Nevi Estimated Size | within three weeks after surgery
  Nevi Estimated Size (centimeters)

SECONDARY OUTCOMES:
post-operative complications depending on the initial size of the naevus | assessed within 6 months after surgery
  post-operative complications depending on the initial size of the naevus : percentage of complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CAPTIER, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC